CLINICAL TRIAL: NCT02721095
Title: Efficacy of KCl Plus 0.9%NaCl Compare With KCl Plus 0.45%NaCl for Correction of Hypokalemia in Hospitalized Patients
Brief Title: Efficacy of KCl Plus 0.9%NaCl Compare With KCl Plus 0.45%NaCl
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMK1981
Record Dates: First submitted 2015-05-25; First posted 2016-03-28 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Hypokalemia
MeSH Terms: conditions — Hypokalemia | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9%NaCl (Experimental): KCl plus 0.9%NaCl
  Interventions: Other: KCl plus 0.9%NaCl
- 0.45%NaCl (Active Comparator): KCl plus 0.45%NaCl
  Interventions: Other: KCl plus 0.45%NaCl

INTERVENTIONS:
Other: KCl plus 0.9%NaCl — comparison of KCl plus 0.9%NaCl and KCl plus 0.45%NaCl for correction of hypokalemia
  Arms: 0.9%NaCl
Other: KCl plus 0.45%NaCl — comparison of KCl plus 0.9%NaCl and KCl plus 0.45%NaCl for correction of hypokalemia
  Arms: 0.45%NaCl

SUMMARY:
evaluate efficacy and safety of IV administration of potassium chloride (KCl) plus 0.9%NaCl compare with KCl plus half-strength normal saline solution (0.45%NaCl) in correcting hypokalemia

DETAILED DESCRIPTION:
Hypokalemia is frequently encountered in hospitalized patients. Intravenous (IV) potassium repletion with saline is preferred used for initial therapy. However, administration of normal saline (0.9%NaCl) usually provokes sodium and potassium diuresis, thus, it might delay reversal of the hypokalemia.

Object of this study : to evaluate efficacy and safety of IV administration of potassium chloride (KCl) plus 0.9%NaCl compare with KCl plus half-strength normal saline solution (0.45%NaCl) in correcting hypokalemia.

ELIGIBILITY:
Inclusion Criteria:

* Serum K+ 2.5-3.49 mmol/L
* No life threatening condition from hypokalemia

Exclusion Criteria:

* Pregnancy
* Volume overload, heart failure
* Hypotension
* Acute kidney injury
* Dysnatremia
* K+ shift
* Salt wasting nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with normal serum K as assessed by serum electrolyte | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yaowana Thanapat, MD, Principal Investigator — Instituitional review board royal thai army medical department
Locations (1):
- Phramonkutklao Hospital, Bangkok, Thailand